CLINICAL TRIAL: NCT01912508
Title: Preterm Labor Prediction by Cervical Contour in Ultrasound
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: MMC-12-0152CTIL
Record Dates: First submitted 2013-07-29; First posted 2013-07-31 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-08

CONDITIONS: Preterm Labor
Keywords: cervical length; cervical curvature
MeSH Terms: conditions — Obstetric Labor, Premature

STUDY DESIGN:
Observational Model: Case-Control

GROUPS / COHORTS (2):
- preterm labor: pregnant women with signs of preterm labor: uterine contractions or cervical shortening
- control: pregnant women with no signs or symptoms of preterm labor

SUMMARY:
Cervical length is a already known predictor for preterm labor. In this study the investigators want to examining the hypothesis that cervical curvature is also a predictor for preterm labor and that moderate transducer pressure influence cervical length.

study population: 200 consecutive pregnant women between 14-34w, visiting in the ultrasound unit ether for routine screening or because of preterm labor.

During their examination cervical length and curvature measurements will be taken. Another measurement will be taken after applying moderate cervical pressure.

The investigators will compere cervical contour and pressure influence between groups and according to cervical length Demographic data will be taken at the time of recruitment and pregnancy outcome measures in a later telephone interview.

ELIGIBILITY:
Inclusion Criteria:

* pregnancy

Exclusion Criteria:

* cervical cerclage
* pre term rupture on membrane in current pregnancy
* unknown dating of pregnancy

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: pregnant women 14-34w
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2013-08; Primary Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
cervical curvature | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Meir hospital, Kfar Saba, Israel